CLINICAL TRIAL: NCT06126627
Title: Neurobiological and Psychobiological Signatures of Vocal Effort in Early Career Teachers
Brief Title: Brain and Voice Signatures in Teachers
Acronym: BRAVO1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Maria Dietrich, Research Associate, University Hospital, Bonn
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R01DC018026 (NIH)
Record Dates: First submitted 2023-10-19; First posted 2023-11-13 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Voice Disorders; Voice Fatigue
Keywords: voice disorders; vocal fatigue; occupational voice disorders; stress reactivity; vocal control; laryngeal motor cortex; teachers; speech motor control; voice motor control
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teachers/student teachers with vocal fatigue (Experimental): Teachers/student teachers with vocal fatigue based on Vocal Fatigue Index (VFI, German). Pre-Screening and Screening. Experiment 1: MRI with MRI-compatible surface electrodes on the neck and audio recordings during MRI with and without stress induction. Prior to MRI, questionnaires on voice, personality, and stress and practice oft the tasks. During experiment, collection of saliva samples (before, during, and after MRI). During MRI, multiple subjective ratings of emotional state by the participants. Experiment 2 (approximately 2 weeks later): Speech tasks with surface electromyographic sensors applied to the neck with concurrent audio recordings. Prior to the experiment questionnaires on voice and practice of tasks. Subjective ratings of vocal and cognitive effort during the experiment by the participants.
  Interventions: Behavioral: Stress induction
- Control group (Active Comparator): Control participants without vocal fatigue based on Vocal Fatigue Index (VFI, German). Same experimental procedures as in arm 1.
  Interventions: Behavioral: Stress induction

INTERVENTIONS:
Behavioral: Stress induction — Induction of anticipatory stress to compare voice and speech control and production with and without exposure to stress.

SUMMARY:
Primary muscle tension dysphonia voice disorder with symptoms of vocal strain and vocal fatigue is common and can have a significant negative impact on quality of Life. Yet, primary muscle tension dysphonia's causes are unknown precluding precise diagnostic classification. Stress and personality are thought to play a role and thus, the project aims to determine the practical and clinical effect of stress on the control of voice and speech in the brain. Participants are female early career teachers and student teachers with symptoms of vocal fatigue, as well as control participants without vocal fatigue, who perform speech tasks on two different occasions. Neural (imaging of brain), psychobiological (saliva, personality), and voice and speech (muscle activity of voice muscles on the neck with surface sensors, audio recordings) data will compare reactivity patterns of teachers who are stressresponders with those who are nonresponders as well as control participants. The central hypothesis is that voice box stress responders have heightened emotion-motor activations involving the emotional voice production pathway, which correlate with changes in voice muscle activity in the anterior neck. The results will provide fundamentally missing data in our understanding of the role of stress in vocal complaints and will yield new insights about the neural underpinnings of primary muscle tension dysphonia. The study findings will have a significant impact on how clinicians identify so-called laryngoresponders to help them prevent voice disorders.

ELIGIBILITY:
Inclusion Criteria:

Teachers (max. 10 years full-time) or student teachers in good health between 21 and 39 years with symptoms of vocal fatigue.

Control participants in good health between 21 and 39 years without symptoms of vocal fatigue.

Exclusion Criteria:

* Lefthandedness
* Smoking (past 5 years)
* Known changes of the vocal folds (e.g., vocal fold nodules), vocal fold paralysis, surgeries on the larynx or thryoid or current organic or neurological changes of the vocal folds or vocal function per videoendoscopy and -stroboscopy of the larynx
* History of voice therapy
* Hoarseness
* Respiratory illness, allergies (respiratory, silver), reflux or asthma at time of participation
* Hearing disorder or hearing aids
* Psychological, neurological or endocrinological disorders
* Psychotropic or steorid medications
* Body mass index > 30
* Indications against MRI such as metail parts in or on the body (e.g., permanent dental prostheses or braces, screws, prostheses, piercings or large tattoos
* Nearsightedness > -5 diopters, if only glasses are worn
* Claustrophobia
* Pregnancy

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Vocal fatigue | through study completion, an average of 1 month
  Raw scores, Vocal Fatigue Index, VFI Factor 1
BOLD MRI area 4p | through study completion, an average of 1 month
  MRI activation in regions of interest (BOLD area 4p in mean %) as a function of speech tasks with and without stress induction
Salivary cortisol | through study completion, an average of 1 month
  Salivary cortisol (nmol/L) to determine stressresponders and nonresponders
Suprahyoid muscle activity | through study completion, an average of 1 month
  Suprahyoid muscle activity (RMS)
Infrahyoid muscle activity | through study completion, an average of 1 month
  Infrahyoid muscle activity (RMS)
Personality, Social Potency | through study completion, an average of 1 month
  Personality trait Social Potency (T-scores, Multidimensional Personality Questionnaire, MPQ)
Personality, Stress Reaction | through study completion, an average of 1 month
  Personality trait Stress Reaction (T-scores, Multidimensional Personality Questionnaire, MPQ)
Personality, social anxiety | through study completion, an average of 1 month
  Personality trait social anxiety (T-scores, Liebowitz Social Anxiety Scale, LSAS-fear)

SECONDARY OUTCOMES:
Vocal fatigue | through study completion, an average of 1 month
  Raw scores, Vocal Fatigue Index, VFI Factor 2 and 3
Voice quality of life | through study completion, an average of 1 month
  Raw data, Voice Handicap Index, VHI
Vocal tract discomfort | through study completion, an average of 1 month
  Raw data, Vocal Tract Discomfort Scale, VTD
Informal questionnaire on vocal health | through study completion, an average of 1 month
  Raw data informal questionnaire on vocal health
BOLD MRI SMA | through study completion, an average of 1 month
  MRI activation in regions of interest (BOLD area SMA in mean %) as a function of speech tasks with and without stress induction
BOLD MRI ACC | through study completion, an average of 1 month
  MRI activation in regions of interest (BOLD area ACC in mean %) as a function of speech tasks with and without stress induction
BOLD MRI MCC | through study completion, an average of 1 month
  MRI activation in regions of interest (BOLD area MCC in mean %) as a function of speech tasks with and without stress induction
BOLD MRI Amygdala | through study completion, an average of 1 month
  MRI activation in regions of interest (BOLD area Amygdala in mean %) as a function of speech tasks with and without stress induction
BOLD MRI PAG | through study completion, an average of 1 month
  MRI activation in regions of interest (BOLD area PAG in mean %) as a function of speech tasks with and without stress induction
Personality, Wellbeing | through study completion, an average of 1 month
  Personality trait Wellbeing (T-scores, Multidimensional Personality Questionnaire, MPQ)
Personality, Social Closeness | through study completion, an average of 1 month
  Personality trait Social Closeness (T-scores, Multidimensional Personality Questionnaire, MPQ)
Personality, social anxiety | through study completion, an average of 1 month
  Personality trait social anxiety (T-scores, Liebowitz Social Anxiety Scale, LSAS-total)
Personality, self-esteem | through study completion, an average of 1 month
  Personality self-esteem (raw data, Rosenberg self-esteem scale)
Behavioral inhibition and exhibition | through study completion, an average of 1 month
  Behavioral inhibition and exhibition (raw data, BIS/BAS scales, BIS subscale)
Chronic Stress | through study completion, an average of 1 month
  Chronic stress (T-scores, Trier Inventory of Chronic Stress, TICS)
Handedness | through study completion, an average of 1 month
  Handedness (raw data, Edinburgh Handedness Inventory, EHI)
State positive and negative affect | through study completion, an average of 1 month
  State positive and negative affect (raw data, Positive and Negative Affect Schedule, PANAS)
Voice quality, relative fundamental frequency | through study completion, an average of 1 month
  Voice quality, relative fundamental frequency (relative fundamental frequency, RFF in semitones [ST])
Voice quality, cepstral-spectral analysis | through study completion, an average of 1 month
  Voice quality, cepstral-spectral analysis (cepstral peak prominence in dB)
Perceived vocal effort | through study completion, an average of 1 month
  Perceived vocal effort (raw data, BORG-CR-10)
Cognitive effort | through study completion, an average of 1 month
  Cognitive effort (raw data, NASA-TLX)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dietrich, PhD, Principal Investigator — University Hospital, Bonn
Locations (1):
- University Hospital Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Yes
The raw data, on which the conclusions are based, will be shared by the authors without any inadmissible caveats starting 6 months post publication with any qualified researcher upon request.